CLINICAL TRIAL: NCT05350722
Title: Single-dose Preoperative Partial Breast Irradiation in Low-risk Breast Cancer Patients
Acronym: ABLATIVE-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Principal Investigator, Desiree H.J.G.D. van den Bongard, MD Ph, MD, PhD, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL77000.029.21
Record Dates: First submitted 2022-03-14; First posted 2022-04-28 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
Keywords: Low-risk breast cancer; Early stage breast cancer; Pre-operative radiotherapy; Partial breast irradiation; Pre-operative single dose radiation; pathologic complete response; cosmetic outcome; survival; toxicity; quality of life; neo-adjuvant radiotherapy; oncological outcomes
MeSH Terms: conditions — Breast Neoplasms; Pathologic Complete Response

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pre-operative single dose partial breast irradiation (Experimental)
  Interventions: Radiation: Single dose ablative radiotherapy

INTERVENTIONS:
Radiation: Single dose ablative radiotherapy — Patients will receive a single dose of 20Gy/15Gy on the gross tumor volume and clinical tumor volume respectively, in the context of pre-operative partial breast irradiation

SUMMARY:
In this ABLATIVE-2 trial, low-risk breast cancer patients will be treated with MRI-guided single dose preoperative partial breast radiotherapy to assess the rate of pathologic complete response after an interval of six to twelve months between radiotherapy and surgery. Response monitoring will be assessed using MRI and markers in blood and tumor tissue to enable prediction of pathologic response.

DETAILED DESCRIPTION:
Patients will receive single-dose preoperative radiotherapy followed by breast conserving surgery (BCS) at 12 months after radiotherapy, as long as follow-up MRI scans show a complete radiologic response. In case of incomplete radiologic response, BCS will be performed at 6 months after radiotherapy. BCS is performed earlier when progressive disease is found on MRI. In the follow-up period between radiotherapy and surgery, tumor response will be monitored using MRI every 3 months. After surgery, patients will be followed up until 10 years after radiotherapy treatment to assess oncological outcomes, toxicity, cosmetic outcome and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* WHO performance scale ≤2.
* Females at least 50 years of age with unifocal cT1N0 breast cancer on mammography, ultrasound and MRI.

  * Patients with an indication for chemotherapy or HER2-targeted therapy according to Dutch National Oncoline Guidelines or own hospital protocols are not eligible. Patients with an indication for endocrine therapy are eligible.
  * Tumor size as assessed on MRI.
* On tumor biopsy:

  * Bloom-Richardson grade 1 or 2.
  * Non-lobular invasive histological type carcinoma.
  * LCIS or (non-extensive) DCIS is accepted.
  * ER positive tumor receptor.
  * HER2 negative tumor.
* Tumor-negative sentinel node (excluding isolated tumor cells).
* Adequate communication and understanding skills of the Dutch language.

Exclusion Criteria:

* Legal incapacity.
* BRCA1, BRCA2 or CHEK2 gene mutation.
* Distant metastasis.
* Previous history of breast cancer or DCIS.
* Other type of malignancy within 5 years before breast cancer diagnosis. Patients with adequately treated malignancy longer than 5 years before breast cancer diagnosis are eligible for inclusion.
* For adequately treated carcinoma in situ of the cervix or basal cell carcinoma of the skin no specific time span to breast cancer diagnosis is required for inclusion.
* Collagen synthesis disease.
* Signs of extensive DCIS component on histological biopsy or on imaging (e.g. no extensive calcifications on mammography).
* Invasive lobular carcinoma.
* MRI absolute contraindications as defined by the Department of Radiology.
* Nodal involvement with cytological or histological confirmation.
* Indication for treatment with (neo-)adjuvant chemotherapy.
* Non-feasible dosimetric RT plan.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2037-12 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response | 12 months after radiotherapy
  pCR is defined as the absence of residual invasive cancer on resected breast specimen

SECONDARY OUTCOMES:
Radiologic complete response | at baseline, 2 weeks, 3, 6, 9, and 12 months after radiotherapy
  Radiologic complete response (rCR) is defined as complete absence of pathologic contrast enhancement in the original tumor bed and complete absence of pathologic ADC (apparent diffusion coefficient) reduction in the original tumor bed. rCR is reported according to the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 guidelines.
Treatment-related adverse events | at baseline, 2 weeks, 3, 6, 9, 12 months, 2, 3, 4, 5, 6, 8 and 10 years after radiotherapy
  Number of participants with treatment-related adverse events as assessed by the Common Terminology Criteria Adverse Events version 5.0
Patient quality of life | at baseline, 2 weeks, 3, 6, 9, 12 months, 2, 3, 4, 5, 6, 8 and 10 years after radiotherapy
  PROMs are assessed using the European Organization for Research and Treatment of Cancer core-30 quality of life questionnaire (EORTC QLQ-C30)
Breast cancer specific quality of life | at baseline, 2 weeks, 3, 6, 9, 12 months, 2, 3, 4, 5, 6, 8 and 10 years after radiotherapy
  PROMs are assessed using the European Organization for Research and Treatment of Cancer breast cancer-specific quality of life questionnaire (EORTC QLQ-BR23)
Patient distress | at baseline, 2 weeks, 3, 6, 9, 12 months, 2, 3, 4, 5, 6, 8 and 10 years after radiotherapy
  PROMs are assessed using the Hospital Anxiety and Depression Scale (HADS) questionnaire
Physician reported cosmetic outcome | at baseline, 2 weeks, 3, 6, 9, 12 months, 2, 3, 4, 5, 6, 8 and 10 years after radiotherapy
  Cosmetic outcome is assessed by the physician using a questionnaire
Patient reported cosmetic outcome | at baseline, 2 weeks, 3, 6, 9, 12 months, 2, 3, 4, 5, 6, 8 and 10 years after radiotherapy
  Cosmetic outcome is assessed by the patient using the BREAST-Q questionnaire. .
Objective cosmetic outcome | at baseline, 2 weeks, 3, 6, 9, 12 months, 2, 3, 4, 5, 6, 8 and 10 years after radiotherapy
  Cosmetic outcome is assessed objectively using images captured using the VECTRA XT 3D-imaging system. This three-dimensional surface-imaging system uses stereophotogrammetry to estimate x, y, z coordinates of the imaged surface. These coordinates will be used to calculate the volume-shape-symmetry measure.
Local, regional and distant relapse rates | Day of radiotherapy till end of follow-up of 10 years
  A local recurrence is defined as disease occurrence in the ipsilateral breast. A regional recurrence is defined as nodal occurrence in the ipsilateral axilla, internal mammary, infraclavicular or supraclavicular region. A distant metastasis defined as disease occurrence in the contralateral breast or contralateral breast nodal region or another organ than breast involvement.
Overall survival | Day of radiotherapy till end of follow-up of 10 years
  Overall survival will be calculated from the date of the radiotherapy treatment until the time of breast-cancer related death or breast-cancer unrelated death.
Radiotherapy-associated immune response markers | 12 months after radiotherapy
  Immune response markers as CD3, CD4, CD8 and FOXP3 will be assessed in tumor tissue after surgery.
Radiotherapy-associated biomarkers | at baseline, 2 weeks, 3, 6, 9, and 12 months after radiotherapy
  ctDNA will be assessed in blood samples taken between radiotherapy and surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Desirée van den Bongard, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (7):
- GenesisCare, Sydney, Australia
- Netherlands (6):
  - Flevoziekenhuis, Almere Stad
  - Ziekenhuis Amstelland, Amstelveen
  - Amsterdam UMC, Amsterdam
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Radboud UMC, Nijmegen
  - Zaans Medisch Centrum, Zaandam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Civil YA, Oei AL, Duvivier KM, Bijker N, Meijnen P, Donkers L, Verheijen S, van Kesteren Z, Palacios MA, Schijf LJ, Barbe E, Konings IRHM, -van der Houven van Oordt CWM, Westhoff PG, Meijer HJM, Diepenhorst GMP, Thijssen V, Mouliere F, Slotman BJ, van der Velde S, van den Bongard HJGD. Prediction of pathologic complete response after single-dose MR-guided partial breast irradiation in low-risk breast cancer patients: the ABLATIVE-2 trial-a study protocol. BMC Cancer. 2023 May 9;23(1):419. doi: 10.1186/s12885-023-10910-6. PMID 37161377